CLINICAL TRIAL: NCT02466360
Title: What Are the Brakes and Levers of Physical Activity Practice for Patients With Chronic Lower Back Pain : a Qualitative Study
Brief Title: What Are the Brakes and Levers of Physical Activity Practice for Patients With Chronic Lower Back Pain?
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Université Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0237
Record Dates: First submitted 2015-06-05; First posted 2015-06-09 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Non-specific Chronic Lower Back Pain
Keywords: Non-specific chronic lower back pain; Physical activity; Self-exercises; Brakes; Levers; Adhesion; Self-care
MeSH Terms: conditions — Motor Activity; Tissue Adhesions | interventions — Focus Groups

STUDY DESIGN:
Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- chronic lower back pain
  Interventions: Behavioral: Back Belief questionnaire; Behavioral: QUEBEC scale; Behavioral: Fear Avoidance beliefs questionnaire; Behavioral: Visual analog scale; Behavioral: individual interviews; Behavioral: Focus groups

INTERVENTIONS:
Behavioral: Back Belief questionnaire
Behavioral: QUEBEC scale
Behavioral: Fear Avoidance beliefs questionnaire
Behavioral: Visual analog scale
Behavioral: individual interviews
Behavioral: Focus groups

SUMMARY:
Non-specific chronic lower back pain is a common pathology which is a real public health problem. Around 84% of the population could have non-specific chronic lower back pain at least once in their lives and 8% of that non-specific lower back pain could become chronical (pain that would last at least 3 months). This proportion of patients represents 85% of the costs related to this pathology.

Physical activity practice is involved in medical care for plenty of chronical diseases and particularly for chronic lower back pain. In 2003, World Health Organization pointed out the poor adhesion of patients with chronical diseases to medical prescriptions and the after-effects it could have on illness evolution. Therefore, adhesion to physical activity practice for patients with chronic lower back pain is one of the most challenging matters for medical teams.

The aim of this study was to identify the brakes and levers of physical activity practice for these patients. Sixteen individual interviews and four focus groups have been carried out on patients with chronic lower back pain who were taken care of either by a rachis functional restoration program or by primary care.

DETAILED DESCRIPTION:
Non-specific chronic lower back pain is a common pathology which is a real public health problem. Around 84% of the population could have non-specific chronic lower back pain at least once in their lives and 8% of that non-specific lower back pain could become chronical (pain that would last at least 3 months). This proportion of patients represents 85% of the costs related to this pathology.

Physical activity practice is involved in medical care for plenty of chronical diseases and particularly for chronic lower back pain. In 2003, World Health Organization pointed out the poor adhesion of patients with chronical diseases to medical prescriptions and the after-effects it could have on illness evolution. Therefore, adhesion to physical activity practice for patients with chronic lower back pain is one of the most challenging matters for medical teams.

The aim of this study was to identify the brakes and levers of physical activity practice for these patients. Sixteen individual interviews and four focus groups have been carried out on patients with chronic lower back pain who were taken care of either by a rachis functional restoration program or by primary care.

ELIGIBILITY:
Inclusion Criteria:

* Male or female who are at least 18 years old
* Patients with non-specific chronic lower back pain

Exclusion Criteria:

* Mental or physical disabilities incompatible with focus groups/individual interviews and filling out questionnaires.
* Inability to understand or speak French properly
* Symptomatic lower back pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with chronic lower back pain
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2012-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Individual interviews | at day 1
  patients with non-specific chronic lower back pain explain directly to their doctors what is preventing them from having physical activity

SECONDARY OUTCOMES:
questions about their lower back pain and physical activity | at day 1
Back Belief questionnaire | at day 1
  - Back Belief questionnaire that evaluates patients' knowledge about lower back pain
QUEBEC scale | at day 1
  - QUEBEC scale that evaluates the impact of lower back pain on the daily lives of patients
Fear Avoidance Beliefs questionnaire | at day 1
  - Fear Avoidance Beliefs questionnaire that evaluates fears and beliefs about the disease
Visual Analog Scale | at day 1
  Visual Analog Scale that evaluates pain

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel COUDEYRE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France